CLINICAL TRIAL: NCT06289036
Title: Predicting Prognosis in Subacute Ischemic Stroke Through Brain Perfusion and Collateral Circulation With Multimodal Imaging
Brief Title: Prognosis in Subacute Ischemic Stroke Using Multimodal Imaging
Status: Completed | Type: Observational
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Zhiyuan Shen, MD, The First Hospital of Hebei Medical University
Other Study IDs: H2020206632
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: The Levels of Cerebral Perfusion and Collateral Circulation in Patients With Subacute Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- favorable prognosis: modified Rankin scale (mRS) ≤ 2
- poor prognosis: modified Rankin scale (mRS) > 2

SUMMARY:
We enrolled patients with subacute IS, associated with moderate-to-severe stenosis of the unilateral cervical internal carotid artery, who underwent 4D ASL. Perfusion levels and collateral circulation were compared between groups with favorable prognosis (modified Rankin scale [mRS] ≤ 2) and poor prognosis (mRS > 2).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed unilateral internal carotid artery/MCA atherosclerotic stenosis/occlusion with a stenosis degree > 50% verified through computed tomography angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA).
2. Presence of IS or transient ischemic attack (TIA) symptoms in the circulating blood supply area within the preceding 48 h.
3. Asymptomatic patients with no history of IS or TIA in the past 6 months.
4. Performance of 4D ASL tests during hospitalization.

Exclusion Criteria:

1. Moderate-to-severe stenosis/occlusion of the contralateral internal carotid artery/middle cerebral arteries.
2. Age ≤ 18 years old.
3. Cardioembolic cerebral infarction.
4. Moyamoya disease.
5. Combined or previous cerebral hemorrhage or subarachnoid hemorrhage
6. History of previous cerebral infarction.
7. Claustrophobia or the presence of intracranial metal implants, cochlear implants, or pacemakers.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with moderate-to-severe stenosis/occlusion of the MCA or carotid artery admitted to the First Hospital of Hebei Medical University between July 2022 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale（mRS） score after 3 months of onset | 3 months
  mRS scores range from 0 to 6, where 0 indicates no symptoms, 3 indicates moderate disability, 4 indicates moderately severe disability, 5 indicates severe disability, and 6 indicates death. Patients were categorized into a good prognosis group (mRS ≤ 2) and a poor prognosis group (mRS > 2).

CONTACTS AND LOCATIONS:
Overall Officials: Shujuan Tian, MD, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No